CLINICAL TRIAL: NCT06619769
Title: eSense-Cancer: Adapting an Online Intervention for Sexual Health Concerns to Gynecologic Cancer
Acronym: eSense-Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Xavier University of Louisiana. (Other)
Responsible Party: Principal Investigator, Lori Brotto, Professor, University of British Columbia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H22-02043
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-02

CONDITIONS: Gynecologic Cancers
Keywords: behavioural intervention; mindfulness based therapy; cognitive behavioural therapy; digital health; eHealth

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either the cognitive-behavioural- or mindfulness-based arm of a digital therapeutic known as eSense-Cancer. Participants will also be randomly assigned to a condition that does or does not include support from a treatment navigator - a non-expert study team member to provide support throughout the treatment. Therefore there will be four groups to be compared:
  * Cognitive-behavioural therapy + navigator support
  * Cognitive-behavioural therapy + no navigator support
  * Mindfulness-based therapy + navigator support
  * Mindfulness-based therapy + no navigator support
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CBT - Navigator (Active Comparator): Participants will complete the CBT arm of eSense with support from a treatment "navigator"
  Interventions: Behavioral: eSense-Cancer CBT: an online cognitive-behavioural therapy based intervention for sexual health concerns after gynecologic cancer; Behavioral: Navigator support for eSense-Cancer
- CBT - No navigator (Active Comparator): Participants will complete the CBT arm of eSense without support from a treatment "navigator"
  Interventions: Behavioral: eSense-Cancer CBT: an online cognitive-behavioural therapy based intervention for sexual health concerns after gynecologic cancer
- MBT - Navigator (Active Comparator): Participants will complete the MBT arm of eSense with support from a treatment "navigator"
  Interventions: Behavioral: Navigator support for eSense-Cancer; Behavioral: Behavioral: eSense-Cancer MBT: an online cognitive-behavioural therapy based intervention for sexual health concerns after gynecologic cancer
- MBT - No navigator (Active Comparator): Participants will complete the MBT arm of eSense without support from a treatment "navigator"
  Interventions: Behavioral: Behavioral: eSense-Cancer MBT: an online cognitive-behavioural therapy based intervention for sexual health concerns after gynecologic cancer

INTERVENTIONS:
Behavioral: eSense-Cancer CBT: an online cognitive-behavioural therapy based intervention for sexual health concerns after gynecologic cancer — eSense-Cancer CBT is an online, cognitive behavioural therapy based intervention for sexual health concerns after gynecologic cancer. eSense-Cancer CBT contains 8 modules and is intended to be completed over 8-16 weeks. It contains theoretical content, case-based learning, and at-home exercises.
  Arms: CBT - Navigator; CBT - No navigator
Behavioral: Navigator support for eSense-Cancer — The eSense digital health tool has been previously tested alongside the support of treatment navigators - trained undergraduate students, not licensed therapists, who provide encouragement and answer any questions users may have as they work through eSense.
  Arms: CBT - Navigator; MBT - Navigator
Behavioral: Behavioral: eSense-Cancer MBT: an online cognitive-behavioural therapy based intervention for sexual health concerns after gynecologic cancer — eSense-Cancer MBT is an online, mindfulness-based therapy based intervention for sexual health concerns after gynecologic cancer. eSense-Cancer MBT contains 8 modules and is intended to be completed over 8-16 weeks. It contains theoretical content, case-based learning, and at-home exercises.
  Arms: MBT - Navigator; MBT - No navigator

SUMMARY:
Sexual health is a vital component of gynecologic cancer treatment and survivorship. Unfortunately, most gynecologic cancer survivors lack sufficient information about the impact of cancer on sexual health and treatment opportunities. This research aims to assess how well an adapted online health intervention meets the sexual health needs of gynecologic cancer survivors and to test the efficacy of the new platform. If successful, eSense-Cancer may increase access to treatment for gynecologic cancer survivors, including those living in remote areas or facing other accessibility barriers. It may also fill healthcare gaps for survivors of varying ethnicity, sexual orientation, socioeconomic status, and gender.

DETAILED DESCRIPTION:
Once participants have consented to participate in the study, they will complete baseline questionnaires, then undergo a 4-week waiting period. After this 4 week waiting period, they will complete a second baseline questionnaire, and then be randomized to one of four arms:

* CBT with navigator support (n=15)
* CBT with no navigator support (n=15)
* MBT with navigator support (n=15)
* MBT with no navigator support (n=15)

Participants will receive an online link to complete the questionnaires consisting of demographics, primary outcomes (sexual distress; FSDS-R, and sexual function; PROMIS SexFS measure adapted for cancer survivors). For those in the navigator support arms, before beginning the eSense-Cancer modules, participants will have an initial 15-30 minute conversation via the UBC-hosted version of Zoom with their assigned navigator, who will explain their role.

Following this meeting, participants will gain access to the CBT or MBT arm of eSense-Cancer and receive an individualized link to access eSense-Cancer. They will work through one module weekly/biweekly (on their own time) and complete the related exercise during that week. This process should take 8-16 weeks. After each module, they will complete a questionnaire to assess usability of the module just completed.

For those in the navigator arms, when participants complete a module, they will fill out their calendar preferences to find a day and time to meet with their navigator over the next week. The navigator will receive an automatic email when their assigned participant has finished a module. If a week has passed and participants have not scheduled a time to meet with their navigator, the navigator will email the participant to schedule their meeting. These meetings will entail 2-3 minutes of general introduction, 10-15 minutes to check in on any eSense-Cancer-related concerns or questions that arose over the week, and 2-3 minutes to close and schedule their next session, for a total of 15-25 minutes.

Navigators will be current or graduated psychology undergraduate students with a GPA of 3.5, coursework or experience with research methods/clinical psychology/human sexuality. Navigators must be available to complete training and commit a minimum of a year to the project. As a licensed clinical psychologist, Dr. Brotto will interview potential navigators to assess their interpersonal skills, ability to listen empathetically, and comfort in discussing sexual issues. Navigators will receive training from co-investigator, Dr. Kyle Stephenson and other study team members to minimize inter-navigator variation. Navigators will have access to both treatment arms to familiarize themselves with eSense-Cancer content. They can choose whether they want to navigate participants in the CBT or MBT arms based on their interests. They will also be given a reading list relevant to treating women's sexual concerns.

After participants complete the final eSense-Cancer module, they will fill out a post-treatment set of questionnaires online. Using the evidence-based framework for feasibility testing, the investigators plan to measure the feasibility dimensions of:

* acceptability: how participants reacted to eSense- Cancer
* implementation: whether the program can be delivered online
* practicality: the ability of a small team to deliver the intervention without providing individualized guidance to participants)
* adaptation: whether the various skills and mindfulness exercises could be delivered online and if participants reported engaging with them)
* limited efficacy testing.

Specific measures include (a) global impressions of eSense-Cancer, (b) preliminary clinical outcomes and (c) navigator-related measures (only administered in the navigator arms):

1. . Global impressions of eSense-Cancer: After completing module 8, participants in both arms will be sent a link and asked qualitative questions on their impressions of the intervention
2. Clinical outcomes:

   1. Sexual distress (FSDS-R)
   2. Sexual function (PROMIS SexFS)
3. Navigator-related measures:

   1. Empathy subscale of Barrett-Lennard Relationship Inventory, a valid measure of perceived provider empathy that predicts outcomes in CBT
   2. Perceived navigator effectiveness with the Working Alliance Inventory, Short Form
   3. Amount of time spent with the participant; each navigator will track how long they spend and engage with each of their assigned participants throughout the eight modules.

The investigators will also use a validated measure of treatment acceptance (Treatment Evaluation Inventory), which has been described as the goodness of fit between the intervention and the system from which it is disseminated), including:

1. The number screened who are appropriate based on study inclusion/exclusion criteria, and from that figure, the number that enrolled in the study.
2. The percentage of participants that completed each intervention module and the entire protocol.
3. The percentage of participants lost to follow-up.

Participants will only receive access to one arm of eSense-Cancer, not both given that our goal is to measure and compare the feasibility and effect size of both arms separately.

Participants' treatment compliance will be measured:

* by recording the number of weeks and treatment sections completed
* through eSense website engagement and performance by a user engagement tracking platform (e.g. page views, #visits/sessions, page views/visits, visit duration, unique/returning users
* by a homework completion measure on a Likert scale ranging from [did not attempt] to [completed all assignments] weekly, which navigators will ask participants to complete
* by having participants complete the Homework Rating Scale (HRS) after each module to provide a comprehensive measure of experience with the homework
* by measuring navigator adherence to study guidelines by recording a random 20% of webcam sessions (with participant knowledge and consent) and coding them for compliance using an adherence scale that the investigators have utilized in the past.

The number of individuals who contact the study coordinator and express interest in the study, regardless of their eligibility, will also be recorded.

During the study, women must agree not to change medications known to have sexual side effects unless directed by their treating physician. (Study investigators will collect data on medication use at each assessment point.) Participants will also be encouraged to limit or eliminate internet research on sexual dysfunction during the trial. The post-treatment questionnaire will assess participant compliance with this request. Past research suggests that this request is feasible.

ELIGIBILITY:
Inclusion Criteria:

* self-report a current or history of gynecologic cancer of any subtype
* self-report symptoms of sexual difficulties and score of greater than 11 on the Female Sexual Distress Scale-Revised
* are fluent in English (eSense content is delivered in English)
* have reliable internet access and basic competency in using online platforms (individuals will self-report)
* are available for 8 - 16 weeks and able to complete eSense modules and associated questionnaires
* any gender

Exclusion Criteria:

* have visual impairments or disabilities interfering with reading and ability to interact with online materials
* have poorly managed anxiety or mood disorder (assessed using the degree of life interference evaluation at screening)
* individuals who are in active treatment for their cancer (including radiation, chemotherapy and any planned surgeries).

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
A change in sexual distress (FSDS-R) | Assessed at enrolment (T1), treatment start (T2) and treatment end (T3). Time between T1 and T2: 4 weeks. Time between T2 and T3: 8-16 weeks
  Sexual distress will be measured using the Female Sexual Distress Scale-Revised (FSDS-R). This scale is measured on a scale of 0-52 with higher values representing more distress.
A change in sexual function and satisfaction (PROMIS SexFs) | Assessed at enrolment (T1), treatment start (T2) and treatment end (T3). Time between T1 and T2: 4 weeks. Time between T2 and T3: 8-16 weeks
  The PROMIS SexFS scale will be used to measure sexual function and satisfaction. The scale consists of 14 questions with higher scores indicating greater levels of sexual function and satisfaction. Scores are differentially calculated for those who are sexually active versus not sexually active.

SECONDARY OUTCOMES:
Treatment satisfaction as assessed by the adapted Erectile Dysfunction Inventory of Treatment Satisfaction | Assessed at post-treatment (T3): 8-16 weeks after treatment start
  Adapted Erectile Dysfunction Inventory of Treatment Satisfaction. Scores range from 0-40, with higher scores reflecting higher treatment satisfaction.
Global Impressions of eSense-Cancer | Assessed at post-treatment (T3): 8-16 weeks after treatment start
  Global impressions of the intervention will be assessed by adapting questions developed by previous work on eSense. All questions are free-response.
Usability of each module | Assessed after completion of each module. There are 8 modules total. Each module should be completed in 1-2 weeks.
  11-items regarding impressions and the ease of use of each module in eSense-Cancer. These are in-house developed items. 5 items are qualitative, 6 items are quantitative.
Treatment satisfaction of each module | Assessed after completion of each module. There are 8 modules total. Each module should be completed in 1-2 weeks.
  Face-valid single-item measures, asking participants to rate helpfulness of content covered each week, and ease of reading the content (0-10 scale). Research suggests a cut-off of 6.5/10 on these measures to indicate acceptable utility and clarity of content. Asked after completing each module.

OTHER OUTCOMES:
Treatment compliance: between-module activity completion assessed by Homework Rating Scale-II (moderator) | Assessed after completion of each module. There are 8 modules total. Each module should be completed in 1-2 weeks.
  Participants complete the Homework Rating Scale-II (HRS-II) after each module. Scores can range from 0-48, with higher scores reflecting high levels of between-module activity completion.
Treatment compliance: Participant engagement with website as assessed by user analytics data capturing (moderator) | Collected throughout engagement with the intervention. Collection will stop at post-treatment (8-16 weeks after treatment start)
  eSense-Cancer website engagement assessed by user analytics data (e.g., total duration of time on website). This will provide a measure of participant engagement.
Treatment compliance: Number of weeks in program (moderator) | Assessed at post-treatment (T3) (8-16 weeks after treatment start).
  Recording number of weeks participant took to complete the program.
Treatment compliance: Number of program modules completed (moderator) | Assessed at post-treatment (T3) (8-16 weeks after treatment start)
  Recording number of program modules participants complete.
Perceived navigator empathy (moderator) | Assessed at post-treatment (T3) for those in a navigator support arm (8-16 weeks after treatment start)
  Empathy subscale of the Barrett-Lennard Relationship Inventory. Scores range from -48 to 48, with higher scores reflecting that participants perceive higher levels of empathy in their navigator.
Perceived navigator alliance (moderator) | Assessed at post-treatment (T3) for those in a navigator arm (8-16 weeks after treatment start)
  Perceived navigator alliance with the Working Alliance Inventory, Short Form. Scores range from 12-84, with higher levels reflecting that participants perceive higher levels of working alliance with their navigator.

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Brotto, PhD, RPsych, Principal Investigator — University of British Columbia; Kyle Stephenson, PhD, RPsych, Principal Investigator — Xavier University of Louisiana.
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
We will be providing all IPD that underlie results in a publication. We will provide Analytic Code only in addition to the data and data dictionaries. Other information will be presented in the publications or available upon request from the main author or PI.
Supporting Information: Analytic Code
Time Frame: The data will be made available within 3 months after publication.
Access Criteria: The data will be freely available on the OSF website so no need for requests.

REFERENCES:
- [Background] Barrett-Lennard GT. The Relationship Inventory: A Complete Resource and Guide.
- [Background] Baker TB, Gustafson DH, Shaw B, Hawkins R, Pingree S, Roberts L, Strecher V. Relevance of CONSORT reporting criteria for research on eHealth interventions. Patient Educ Couns. 2010 Dec;81 Suppl:S77-86. doi: 10.1016/j.pec.2010.07.040. Epub 2010 Sep 16. PMID 20843621
- [Background] Derogatis L, Clayton A, Lewis-D'Agostino D, Wunderlich G, Fu Y. Validation of the female sexual distress scale-revised for assessing distress in women with hypoactive sexual desire disorder. J Sex Med. 2008 Feb;5(2):357-64. doi: 10.1111/j.1743-6109.2007.00672.x. Epub 2007 Nov 27. PMID 18042215
- [Background] Kazdin AE. Acceptability of alternative treatments for deviant child behavior. J Appl Behav Anal. 1980 Summer;13(2):259-73. doi: 10.1901/jaba.1980.13-259. PMID 7380752
- [Background] Brotto LA, Stephenson KR, Zippan N. Feasibility of an Online Mindfulness-Based Intervention for Women with Sexual Interest/Arousal Disorder. Mindfulness (N Y). 2022;13(3):647-659. doi: 10.1007/s12671-021-01820-4. Epub 2022 Jan 4. PMID 35035598